CLINICAL TRIAL: NCT03963297
Title: Multicenter Evaluation of the Susceptibility of Enterobacteriaceae and Pseudomonas Aeruginosa to Ceftolozane/Tazobactam Combination
Acronym: GMC-9
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: GMC-9
Record Dates: First submitted 2019-05-15; First posted 2019-05-24 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Antibiotic Resistant Strain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For hospitalized patients who may have a community or nosocomial Gram-negative bacillus infection of the enterobacterial type or P. aeruginosa type, diagnostic specimens are taken by the clinical department and sent to the local microbiology laboratory for investigation, in accordance with standard management. Depending on the location, the samples may be AMLs (Bronchial-Alveolar Washing), PDPs (Protected Distal Sampling), blood culture, ascites, operating room samples or other puncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ceftolozane/tazobactam is a new antibiotic with broad spectrum activity. This molecule is currently one of the most active beta lactams against Pseudomonas aeruginosa and its spectrum of activity also includes enterobacteriaceae producing a broad spectrum beta-lactamase (EBLSE). Ceftolozane/tazobactam is currently marketed for the treatment of complicated intra-abdominal infections and complicated urinary tract infections. These intra-abdominal and urinary infections are mainly caused by enterobacteriaceae (Escherichia coli, Klebsiella pneumoniae) and more rarely by P. aeruginosa. Concerning enterobacteriaceae, French epidemiology reports a prevalence of BLSE of between 10 and 15% in E. coli and 10%-30% in K. pneumoniae.

DETAILED DESCRIPTION:
Currently, the probabilistic treatment of these multi-resistant bacteria involves the use of carbapenems. Unfortunately, the increasing and unreasonable use of carbapenems invariably leads to the spread of even more resistant strains, BHRe (Emerging Highly Resistant Bacteria) including enterobacteriaceae producing carbapenemases. Thus, it is strongly recommended by health authorities to limit the use of carbapenems ("carbapenem savings") by promoting the use of therapeutic alternatives. Ceftolozane/tazobactam is one of those therapeutic alternatives for which an evaluation must be carried out. Currently, in addition to complicated intra-abdominal infections and complicated urinary tract infections, ceftolozane/tazobactam combination is used in clinical practice in gram-negative infections such as upper and lower respiratory infections and bacteremia. In any case, the choice of probabilistic antibiotic therapy must take into account local and regional epidemiological data. However, published data on the in vitro activity of ceftolozane/tazobactam remain limited, particularly in France (only one French epidemiological study on Gram-negative non-fermenting bacillus strains isolated in patients with cystic fibrosis). This study does not take into account in particular multi-resistant enterobacteriaceae producing BLSE for which ceftolozane/tazobactam remains effective (particularly in E. coli and K. pneumoniae).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years old
* Hospitalized patient with community-acquired or nosocomial Gram-negative bacillus infection of enterobacteriaceae or P. aeruginosa type (bacteremia, low respiratory infection, intra-abdominal infection)
* French-speaking patient

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient under the protection of justice
* Refusal to participate in the study
* Patients judged by the investigator as being unable to express their non-opposition to the study
* Urinary localization of the infection to avoid strains responsible for simple colonization. Indeed, the collection of microbiological data (as carried out in this study) makes it difficult to distinguish between real infection and simple colonization. In addition, the impact of early implementation of appropriate therapy on the evolution of infectious disease (mortality, morbidity, etc.) has been clearly demonstrated for serious infections such as bacteremia and respiratory infections, while this impact remains more limited or even insignificant for urinary infections. Hence the desire to exclude isolated strains of urine samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient with community-acquired or nosocomial Gram-negative bacillus infection of enterobacteriaceae or P. aeruginosa type (bacteremia, low respiratory infection, intra-abdominal infection)
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Value of the minimum inhibitory concentration (MIC) | 1 year
  Value of the minimum inhibitory concentration (MIC) obtained for ceftolozane/tazobactam for each strain

SECONDARY OUTCOMES:
Patient History | 1 year
  Clinical profil of patients (yes/no) correlated with resistance or susceptibility of strains to ceftolozane/tazobactam
Number of strains producing ESBL and/or carbapenemase (yes or no) | 1 year
  biochemical tests (ESBL NDP test and/or Carba NP test)
Molecular profil of enterobacteriaceae (produced genes : yes or no) | 1 year
  Molecular test (PCR + sequencing: blaCTX-M, blaTEM, blaSHV)
Molecular profil of pseudomonas aeruginosa (produced genes : yes or no) | 1 year
  Molecular test (PCR + sequencing : blaGES, blaVEB and blaPER)

CONTACTS AND LOCATIONS:
Overall Officials: Alban Le Monnier, Professor, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Castanheira M, Duncan LR, Mendes RE, Sader HS, Shortridge D. Activity of Ceftolozane-Tazobactam against Pseudomonas aeruginosa and Enterobacteriaceae Isolates Collected from Respiratory Tract Specimens of Hospitalized Patients in the United States during 2013 to 2015. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e02125-17. doi: 10.1128/AAC.02125-17. Print 2018 Mar. PMID 29263073
- [Result] Walkty A, Adam H, Baxter M, Lagace-Wiens P, Karlowsky JA, Hoban DJ, Zhanel GG. In vitro activity of ceftolozane/tazobactam versus antimicrobial non-susceptible Pseudomonas aeruginosa clinical isolates including MDR and XDR isolates obtained from across Canada as part of the CANWARD study, 2008-16. J Antimicrob Chemother. 2018 Mar 1;73(3):703-708. doi: 10.1093/jac/dkx468. PMID 29244121
- [Result] Monogue ML, Nicolau DP. Antibacterial activity of ceftolozane/tazobactam alone and in combination with other antimicrobial agents against MDR Pseudomonas aeruginosa. J Antimicrob Chemother. 2018 Apr 1;73(4):942-952. doi: 10.1093/jac/dkx483. PMID 29272436
- [Result] Munita JM, Aitken SL, Miller WR, Perez F, Rosa R, Shimose LA, Lichtenberger PN, Abbo LM, Jain R, Nigo M, Wanger A, Araos R, Tran TT, Adachi J, Rakita R, Shelburne S, Bonomo RA, Arias CA. Multicenter Evaluation of Ceftolozane/Tazobactam for Serious Infections Caused by Carbapenem-Resistant Pseudomonas aeruginosa. Clin Infect Dis. 2017 Jul 1;65(1):158-161. doi: 10.1093/cid/cix014. PMID 28329350
- [Result] Chen M, Zhang M, Huang P, Lin Q, Sun C, Zeng H, Deng Y. Novel beta-lactam/beta-lactamase inhibitors versus alternative antibiotics for the treatment of complicated intra-abdominal infection and complicated urinary tract infection: a meta-analysis of randomized controlled trials. Expert Rev Anti Infect Ther. 2018 Feb;16(2):111-120. doi: 10.1080/14787210.2018.1429912. Epub 2018 Jan 24. PMID 29343141